CLINICAL TRIAL: NCT02573337
Title: A Multi-center, Non-comparative Study to Evaluate the Perception of Facial Expressions Following Correction of Wrinkles and Folds in the Lower Face Using Emervel Classic Lidocaine and Emervel Deep Lidocaine
Brief Title: Perception of Facial Expressions Following Correction of Wrinkles and Folds
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05DF1502
Record Dates: First submitted 2015-10-08; First posted 2015-10-09 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2016-01

CONDITIONS: Wrinkles and Folds in Lower Face

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intradermal injection (Experimental): Emervel Classic Lidocaine and/or Emervel Deep Lidocaine
  Interventions: Device: Emervel Classic Lidocaine; Device: Emervel Deep Lidocaine

INTERVENTIONS:
Device: Emervel Classic Lidocaine — Treatment of wrinkles and folds
Device: Emervel Deep Lidocaine — Treatment of wrinkles and folds

SUMMARY:
The purpose of this study is to evaluate the perception of facial expressions following correction of wrinkles and folds in the lower face using Emervel Classic Lidocaine and Emervel Deep Lidocaine.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* NLFs assessed as moderate of severe using the WSRS
* Intent to undergo optimal correction of both NLFs
* Intent to undergo correction of at least one other wrinkle or fold in the lower face

Exclusion Criteria:

* Subject who presents with a severity of wrinkles or folds that require other treatments, e.g. laser treatment, chemical peeling, to achieve optimal correction
* Subject who presents with severe midface volume loss
* Subject who presents with facial hair, e.g. beard, moustache, in the treatment area
* Woman who is pregnant or breast feeding or plans to become pregnant during the study
* Treatment with chemotherapy, immunosuppressive agents, immunomodulatory therapy (e.g. monoclonal antibodies), systemic or topical (facial) corticosteroids (inhaled corticoids are allowed) within three (3) months before study treatment
* Previous surgery, including aesthetic facial surgical therapy, liposuction or tattoo, in the treatment area
* Previous tissue augmenting therapy or contouring with permanent filler or fat-injection below the zygomatic arch
* Previous tissue augmenting therapy, contouring or revitalisation treatment with non-HA filler, e.g. Calcium Hydroxyapatite (CaHa), or Poly L-Lactic Acid (PLLA), below the zygomatic arch within 24 months before treatment
* Previous tissue augmenting therapy, contouring or revitalisation treatment with non-permanent filler below the zygomatic arch within 12 months before treatment
* Previous tissue revitalisation treatment with neurotoxin below the zygomatic arch within six (6) months before treatment
* Previous tissue revitalisation treatment with laser or light, mesotherapy, chemical peeling or dermabrasion below the zygomatic arch within six (6) months before treatment
* Any medical condition that, in the opinion of the treating investigator, would make the subject unsuitable for inclusion (e.g. a chronic, relapsing or hereditary disease that may interfere with the outcome of the study)

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Treatment impact on facial expressions | 1 month after touch-up treatment
  Perception of naturalness

SECONDARY OUTCOMES:
Safety by assessment of local tolerability | 2 weeks after first treatment
Safety by assessment of Adverse Events | 0-13 months
Treating investigator satisfaction with treatment outcome | 1 month after touch-up
  Questionnaire
Subject satisfaction with treatment outcome | 1 month after touch-up
  Questionnaires
Nasolabial fold severity | Before treatment and 2 weeks after first treatment and 1 month after touch-up
  WSRS photo scale
Aesthetic improvement of lower face | 1 month after touch-up
  GAIS

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Cologne
  - Darmstadt
  - Munich